CLINICAL TRIAL: NCT02871765
Title: The Educational Effectiveness for Atrial Fibrillation Patients Under Warfarin Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 98-3227B
Record Dates: First submitted 2016-08-01; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
Keywords: Patient education; Knowledge; Life distress; Quality of life
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- education group (Experimental): In education group, each subject in the experimental group was taught individually according to investigator's brochure in the outpatient department by researchers. Three months later, participants in the education group received a follow-up phone call in order to clarify any questions related to the brochure. All participants completed posttest at 6-month follow-up.
  Interventions: Other: Patient education related Warfarin
- control group (No Intervention): The control group received the brochure only.

INTERVENTIONS:
Other: Patient education related Warfarin — Patient education related Warfarin: each subject in the experimental group was taught individually according to investigator's brochure in the outpatient department (OPD) by researchers. Three months later, participants received a follow-up phone call in order to clarify any questions related to the brochure. The contents of the brochure consisted of: the purpose of taking Warfarin, side effects, adjustments to daily diet, and precautions (i.e. how to take medication safely, interaction between foods and medicine, prevention and checking of signs and symptoms of bleeding). The control group received the brochure after pretest and routine care only in the OPD. All participants completed posttest at 6-month follow-up.
  Arms: education group

SUMMARY:
The objective of this study is to evaluate an educational program for Atrial Fibrillation patients under Warfarin treatment regarding to patients' knowledge of Warfarin, related life distresses and quality of life.

DETAILED DESCRIPTION:
This is a parallel-group randomized controlled study. Four measurements were (a) knowledge of Warfarin; (b) life distresses caused by Warfarin treatment; and (c) quality of life as primary and secondary endpoint. All participants participated in a face-to-face interview during the pretest and at the 6-month follow-up in the outpatient department (OPD). Each subject in the experimental group was taught face-to-face individually according to investigator's brochure in the OPD by researchers trained in a standardized protocol. The control group received a brochure only.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Atrial Fibrillation by a physician and taking Warfarin as treatment
* 20 years old or older
* clear consciousness for communication
* willingness to participate in research

Exclusion Criteria:

* can not communicate clearly
* without willingness to participate in research

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
knowledge of Warfarin | 6-month follow-up
  There were six questions and the contents were consistent with investigator's brochure used in investigator's research setting. When participants answered questions correctly, or illustrated at least two correct examples for each item, participants received one point; otherwise, participants received no point. The range of scores was 0-6. The higher the score, the better the patient's knowledge of Warfarin was.

SECONDARY OUTCOMES:
life distress | 6-month follow-up
  There were six questions. The most commonly cited things patients suffered from while under Warfarin treatment were included. When participants answered "yes", participants received one point; if participants answered "no", participants received no point. The range of scores was 0-6. A higher score indicated a worse life distresses.
quality of life | 6-month follow-up
  Investigators use SF-36 to measure participants' quality of life.The SF-36 consists of eight scaled scores, including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health,which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: YU-HSIA TSAI, MS,RN, Principal Investigator — Chang Gung University

IPD SHARING:
Plan to Share IPD: Yes
Investigators are going to publish research results.

REFERENCES:
- [Background] Pernod G, Labarere J, Yver J, Satger B, Allenet B, Berremili T, Fontaine M, Franco G, Bosson JL. EDUC'AVK: reduction of oral anticoagulant-related adverse events after patient education: a prospective multicenter open randomized study. J Gen Intern Med. 2008 Sep;23(9):1441-6. doi: 10.1007/s11606-008-0690-1. Epub 2008 Jun 20. PMID 18566863
- [Background] Wofford JL, Wells MD, Singh S. Best strategies for patient education about anticoagulation with warfarin: a systematic review. BMC Health Serv Res. 2008 Feb 14;8:40. doi: 10.1186/1472-6963-8-40. PMID 18275605
- [Background] Casais P, Meschengieser SS, Sanchez-Luceros A, Lazzari MA. Patients' perceptions regarding oral anticoagulation therapy and its effect on quality of life. Curr Med Res Opin. 2005 Jul;21(7):1085-90. doi: 10.1185/030079905X50624. PMID 16004677